CLINICAL TRIAL: NCT02117414
Title: Evera MRI Clinical Study
Brief Title: Confirmatory Clinical Trial of the Evera MRI System for Conditionally-safe MRI Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Evera MRI
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Implantable Defibrillator
Keywords: Magnetic Resonance Imaging (MRI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI Group (Experimental): Subjects randomized to the MRI group will undergo a series of MRI scans at the MRI visit (9-12 weeks post-implant).
  Interventions: Device: MRI scan sequences of the head and chest regions
- Control Group (Sham Comparator): Subjects randomized to the Control group will wait for 1 hour without having a series of MRI scans at the waiting period visit (9-12 weeks post-implant).
  Interventions: Other: Waiting Period Visit

INTERVENTIONS:
Device: MRI scan sequences of the head and chest regions — Non-diagnostic MRI scans
  Arms: MRI Group
Other: Waiting Period Visit — Waiting period time will equate to 1 hour
  Arms: Control Group

SUMMARY:
The purpose of the Evera MRI™ study is to confirm safety and efficacy of the Evera MRI ICD (Implantable cardioverter-defibrillator) System in the clinical MRI (Magnetic Resonance Imaging) environment when subjects receive MRI scans without positioning restrictions (MRI scans may occur anywhere on the body).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are indicated for implantation of an ICD at the time of study enrollment.
* Subjects who are able to undergo a pectoral implant.
* Subjects who are receiving an ICD for the first time.
* Subjects who are able and willing to undergo elective MRI scanning without sedation.
* Subjects who are geographically stable and available for follow-up at the study site for the length of the study.
* Subjects who are at least 18 years of age (or older, if required by local law).

Exclusion Criteria:

* Subjects with a history of significant tricuspid valvular disease .
* Subjects for whom a single dose of 1.0mg dexamethasone sodium phosphate and/or dexamethasone acetate may be contraindicated.
* Subjects who require a legally authorized representative to obtain informed consent.
* Subjects undergoing device upgrades, change-outs, lead extractions, and/or lead or device revisions.
* Subjects with abandoned or capped leads.
* Subjects who require an indicated MRI scan, other than those specifically described in the Evera MRI™ study, before the one-month post-MRI/waiting period follow-up (approximately 4 months post-implant).
* Subjects with a non-MRI compatible device (such as neurostimulators) or material implant (e.g., non-MRI compatible sternal wires, neurostimulators, biostimulators, metals or alloys).
* Subjects with medical conditions that preclude the testing required by the study protocol or limit study participation.
* Subjects who are enrolled or intend to participate in another clinical trial (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during the Evera MRI™ study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.
* Female patient who is pregnant, or of childbearing potential and not on a reliable form of birth control. Women of childbearing potential are required to have a negative pregnancy test within seven (7) days prior to device implant.
* Subjects with exclusion criteria required by local law (e.g., age, breastfeeding).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Gold, MD, PhD, Principal Investigator — Medical University of South Carolina; Emanuel Kanal, MD, FACR, Principal Investigator — University of Pittsburgh Medical Center, USA; Juerg Schwitter, MD, Principal Investigator — University Hospital Lausanne (CHUV), Switzerland; Torsten Sommer, MD, Principal Investigator — German Red Cross Hospital (DRK) Neuwied, Germany
Locations (42):
- United States (25):
  - Central Coast Cardiology, Salinas, California
  - Stanford Hospitals & Clinics, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Orlando Health, Orlando, Florida
  - Prairie Education & Research Cooperative (Springfield IL), Springfield, Illinois
  - Iowa Heart, West Des Moines, Iowa
  - Washington Hospital Center, Washington DC, Maryland
  - DLP Upper Michigan Cardiovascular Associates PC, Marquette, Michigan
  - Park Nicollet Methodist Hospital, Saint Louis Park, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Mid America Heart Institute (MAHI), Kansas City, Missouri
  - HealthCare Partners CCNV, Henderson, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - NYU Langone Medical Center, New York, New York
  - University of North Carolina (UNC) Memorial Hospital, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Centre Hospitalier Régional de la Citadelle, Liège, Belgium
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec
- Hospital Clínico Pontificia Universidad Católica, Santiago, Chile
- Germany (4):
  - Universitätsklinikum Bonn, Bonn
  - Praxisklinik Herz und Gefässe, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena - Friedrich Schiller Universität, Jena
- Queen Mary Hospital, Hong Kong, Hong Kong
- Semmelweis Egyetem AOK, Budapest, Hungary
- Medanta-The Medicity, Gūrgaon, India
- Azienda Ospedaliera SS Annunziata, Taranto, Italy
- HagaZiekenhuis - Locatie Leyweg, The Hague, Netherlands
- Prince Sultan Cardiac Center, Riyadh, Saudi Arabia
- Akademiska Sjukhuset, Uppsala, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Schwitter J, Gold MR, Al Fagih A, Lee S, Peterson M, Ciuffo A, Zhang Y, Kristiansen N, Kanal E, Sommer T; Evera-MRI Study Investigators. Image Quality of Cardiac Magnetic Resonance Imaging in Patients With an Implantable Cardioverter Defibrillator System Designed for the Magnetic Resonance Imaging Environment. Circ Cardiovasc Imaging. 2016 May;9(5):e004025. doi: 10.1161/CIRCIMAGING.115.004025. PMID 27151268
- [Derived] Gold MR, Sommer T, Schwitter J, Al Fagih A, Albert T, Merkely B, Peterson M, Ciuffo A, Lee S, Landborg L, Cerkvenik J, Kanal E; Evera MRI Study Investigators. Full-Body MRI in Patients With an Implantable Cardioverter-Defibrillator: Primary Results of a Randomized Study. J Am Coll Cardiol. 2015 Jun 23;65(24):2581-2588. doi: 10.1016/j.jacc.2015.04.047. Epub 2015 May 14. PMID 25982014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 275 subjects were enrolled (consented) at 42 centers in the Evera MRI study. The first enrollment occurred on April 17, 2014, and the last enrollment occurred on September 11, 2014.
Pre-assignment Details: A successful implant was defined as having received a complete Evera MRI™ Study System (Evera MRI™ DR or VR ICD, one Model 6935M or 6947M lead, and one Model 5076 lead (if DR system)). Eleven subjects did not have an implant attempt and one subject did not have a successful implant. None of these subjects were randomized.
Period: Overall Study
Arm/Group | MRI Group | Control Group
Started | 175 (Subjects randomized to the MRI group.) | 88 (Subjects randomized to the Control group.)
Completed | 160 (Subject followed up at least to the one-month post MRI/Waiting period visit in the MRI group.) | 82 (Subject followed up at least to the one-month post MRI/Waiting period visit in the Control group.)
Not Completed | 15 | 6
Not completed — Death | 5 | 2
Not completed — Withdrawal by Subject | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRI Group | Control Group | Total
Number analyzed (Participants) | 175 | 88 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (13.5) | 60.1 (14.3) | 60.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 22 | 62
  Male | 135 | 66 | 201

OUTCOME MEASURES:

1. Primary Outcome: MRI-related Events
Description: Number of patients free of MRI-related events. Events include MRI-related complications, sustained tachyarrhythmia, and MRI-related loss of pacing ability.
Time Frame: MRI procedure to 1-month post-MRI
Population: A total of 156 subjects underwent an MRI scan at the MRI/waiting period visit; of them 147 were followed through the one month post-MRI visit or later and are included in the analysis.
Measure: Number; unit: Participants free of MRI-related events
Groups:
- MRI Group: All subjects successfully implanted with the Evera MRI Study System who have an MRI scan at the MRI/waiting period visit and have completed their one month post-MRI scan follow-up, (or a later follow-up), or have had an MRI-related event without completion of their one-month post-MRI scan follow-up will be included in the analysis
Arm/Group | MRI Group
Number analyzed (Participants) | 147
Participants free of MRI-related events | 147
Statistical Analysis 1: Comparison: MRI Group; The alternative hypothesis is that the MRI-related event-free rate between the MRI procedure and one month post-MRI is greater than 90%. The null hypothesis will be rejected if the one-sided 97.5% lower confidence bound is greater than 90% or, equivalently, if the p-value is less than 0.025. Assuming type I error rate 0.025, even-free rate under null hypothesis 90% and true even-free rate 0.995, the minimum required sample size is 54 MRI scanned subjects in order to obtain 90% power; Test type: Superiority or Other; p < 0.0001, one-proportion binomial exact test — A priori threshold for statistical significance was 0.025; Percentage = 100, 95% CI 1-sided [lower limit 97.75]

2. Primary Outcome: Ventricular Pacing Capture Threshold (VPCT)
Description: Number of successful patients, where success is defined as not increasing VPCT by more than 0.5V from pre-MRI/waiting to one month post.
Time Frame: Pre-MRI/Waiting Period visit to 1-month post-MRI/Waiting Period visit
Population: To be included in the analysis, subjects in the MRI group must undergo an MRI scan and those in the Control group must complete the MRI/waiting period visit, and all the subjects must have valid VPCT measurements pre-MRI/waiting period and post-MRI/waiting period.
Measure: Number; unit: Successful participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 154 | 81
Successful participants | 154 | 80
Statistical Analysis 1: Comparison: MRI Group vs Control Group; The percentage of subjects who experience a VPCT increase less than or equal to 0.5V from the pre-MRI/waiting period to one month post-MRI/waiting period in the MRI group is greater than that in the Control group minus 10%. H0: % successes MRI group ≤ % successes Control group - 10% HA: % successes MRI group > % successes Control group - 10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; p < 0.0001, Farrington-Manning non-inferiority test — A priori threshold for statistical significance was 0.025; Difference in percentages = 1.2, 95% CI 1-sided [lower limit -3.8]

3. Primary Outcome: Ventricular Sensing Amplitude (R-wave)
Description: Number of successful patients who do not experience a decrease in ventricular sensing amplitude of >50% from the pre-MRI/waiting period to the one month post-MRI/waiting period, or a one month post-MRI/waiting value <3mV accompanied by a decrease of >25% from the pre-MRI/waiting period to the one month post-MRI/waiting period.
Time Frame: Pre-MRI/Waiting Period visit to 1-month post-MRI/Waiting Period visit
Population: Only subjects with measured ventricular sensing amplitude values both pre-MRI/waiting period and post-MRI/waiting period were used in the analysis.
Measure: Number; unit: Successful participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 153 | 82
Successful participants | 152 | 81
Statistical Analysis 1: Comparison: MRI Group vs Control Group; The percentage of subjects who do not experience a significant decrease in ventricular sensing amplitude from the pre-MRI/waiting period to one month post-MRI/waiting period is greater than that in the Control group minus 8%. H0: % successes MRI group ≤ % successes Control group - 8% HA: % successes MRI group > % successes Control group - 8%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 8%; p = 0.0001, Farrington-Manning non-inferiority test — A priori threshold for statistical significance was 0.025; Difference in percentages = 0.6, 95% CI 1-sided [lower limit -4.1]

4. Secondary Outcome: System-related Complications
Description: Number of subjects free of a system-related complication. The system includes the ICD and lead(s) attached to it.
Time Frame: Implant to 4 months post-implant
Population: All subjects who are successfully implanted with the Evera MRI Study System or have an implant attempt will be included in the analysis.
Measure: Number; unit: Successful participants
Groups:
- Implanted Subjects: All subjects who are successfully implanted with the Evera MRI Study System or have an implant attempt will be included in the analysis.
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 264
Successful participants | 254
Statistical Analysis 1: Comparison: Implanted Subjects; The system-related complication-free rate between the implant procedure and the one month post-MRI/waiting period is greater than 80%. H0: p ≤ 0.80 HA: p > 0.80 where p is the system-related complication-free rate between the implant procedure and 120 days (the approximate time of the one month post-MRI/waiting period visit); Test type: Non-Inferiority or Equivalence — The null hypothesis will be rejected if the one-sided 95% log-log transformed lower confidence bound at 120 days post-implant calculated using Kaplan-Meier (K-M) method is greater than 80%; p < 0.0001, Kaplan-Meier method — A priori threshold for statistical significance was 0.05; Complication-free rate = 95.9, 95% CI 1-sided [lower limit 93.0]

5. Secondary Outcome: RV Defibrillation Impedance
Description: Number of subjects whose RV defibrillation impedance at the one-month post-MRI/waiting period visit is between 20 and 100 ohms
Time Frame: 1-month post-MRI/Waiting Period visit
Population: Only randomized subjects with measured RV defibrillation impedance one month post-MRI/waiting period were used in the analysis. The percentages of subjects with an RV defibrillation impedance between 20 and 100 ohms at the one month post-MRI/waiting period visit were calculated.
Measure: Number; unit: Successful participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 145 | 81
Successful participants | 145 | 80
Statistical Analysis 1: Comparison: MRI Group vs Control Group; The percentage of subjects who have a defibrillation impedance between 20 and 100 ohms at the one month post-MRI/waiting period visit in the MRI group is greater than that in the Control group minus 10%. H0: % successes MRI group ≤ % successes Control group - 10% HA: % successes MRI group > % successes Control group - 10% Where % successes means the % of subjects whose defibrillation impedance at the one month post-MRI/waiting period visit is between 20 and 100 ohms; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 10%; p < 0.00001, Farrington-Manning non-inferiority test — A priori threshold for statistical significance was 0.05; Difference in percentages = 1.2, 90% CI 1-sided [lower limit -3.1]

6. Secondary Outcome: Superior Vena Cava (SVC) Defibrillation Impedance
Description: Number of subjects whose SVC defibrillation impedance at the one-month post-MRI/waiting period visit is between 20 and 100 ohms
Time Frame: 1-month post-MRI/Waiting Period visit
Population: Only randomized subjects with measured SVC defibrillation impedance one month post-MRI/waiting period were used in the analysis. The percentages of subjects with an SVC defibrillation impedance between 20 and 100 ohms at the one month post-MRI/waiting period visit were calculated.
Measure: Number; unit: Successful participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 42 | 25
Successful participants | 42 | 25
Statistical Analysis 1: Comparison: MRI Group vs Control Group; The percentage of subjects who have a SVC defibrillation impedance between 20 and 100 ohms at the one month post-MRI/waiting period visit in the MRI group is greater than that in the Control group minus 10%. H0: % successes MRI group ≤ % successes Control group - 10% HA: % successes MRI group > % successes Control group - 10% Where % successes means the % of subjects whose SVC defibrillation impedance at the one month post-MRI/waiting period visit is between 20 and 100 ohms; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 10%; Farrington-Manning non-inferiority test — A priori threshold for statistical significance was 0.05. Because the success rate was 100% in each group, a p-value could not be calculated; Difference in percentages = 0

7. Secondary Outcome: Atrial Pacing Capture Threshold (APCT)
Description: Number of successful patients, where success is defined as not increasing APCT by more than 0.5V from pre-MRI/waiting to one month post.
Time Frame: Pre-MRI/Waiting Period visit to 1-month post-MRI/Waiting Period visit
Population: To be included in the analysis, subjects in the MRI group must undergo an MRI scan and those in the Control group must complete the MRI/waiting period visit, and all the subjects must have valid APCT measurements pre-MRI/waiting period and post-MRI/waiting period.
Measure: Number; unit: Successful participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 75 | 32
Successful participants | 74 | 32
Statistical Analysis 1: Comparison: MRI Group vs Control Group; The percentage of subjects who experience an APCT increase less than or equal to 0.5V from the pre-MRI/waiting period to one month post-MRI/waiting period in the MRI group is greater than that in the Control group minus 10%. H0: % successes MRI group ≤ % successes Control group - 10% HA: % successes MRI group > % successes Control group - 10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 10%; p = 0.006, Farrington-Manning non-inferiority test; Difference in percentages = -1.3, 90% CI 1-sided [lower limit -7.0]

8. Secondary Outcome: Atrial Sensing Amplitude
Description: Number of successful patients, where success is defined as not decreasing atrial sensing amplitude by more than 50% from pre-MRI/waiting to one month post.
Time Frame: MRI/waiting visit to 1-month post-MRI/Waiting visit
Population: Only subjects with measured atrial sensing amplitude values at both the pre-MRI/waiting period and post-MRI/waiting period were used in the analysis.
Measure: Number; unit: Successful participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 76 | 34
Successful participants | 74 | 33
Statistical Analysis 1: Comparison: MRI Group vs Control Group; The percentage of subjects who do not experience a 50% decrease in atrial sensing amplitude from the pre-MRI/waiting period to one month post-MRI/waiting period is greater than that in the Control group minus 10%. H0: % successes MRI group ≤ % successes Control group - 10% HA: % successes MRI group > % successes Control group - 10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 10%; p = 0.005, Farrington-Manning non-inferiority test — A priori threshold for statistical significance was 0.05; Difference in percentages = 0.3, 90% CI 1-sided [lower limit -6.2]

ADVERSE EVENTS:
Time Frame: The 263 randomized subjects averaged 4.5 months of implanted follow-up for a total of 97.6 years of follow-up.
Description: There were 158 adverse events in randomized subjects.
Arm/Group | MRI Group | Control Group
Serious Adverse Events (participants affected / at risk) | 35/175 | 15/88
Other Adverse Events (participants affected / at risk) | 0/175 | 0/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Group (N=175) | Control Group (N=88)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 5 (5) | 5 (6)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 3 (4)
Death (General disorders) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Lead dislodgement (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and Participating Institutions will provide any publication of Study Data generated by PI and/or Participating Institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.